CLINICAL TRIAL: NCT00614874
Title: The Effects of the PPARy Agonist Rosiglitazone on Airway Hyperreactivity
Brief Title: The Use of Rosiglitazone to Treat Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Tammy Wichman, Associate Professor of Medicine, Creighton University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-14592
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2011-09-02 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-09

CONDITIONS: Asthma
Keywords: Asthma; Avandia
MeSH Terms: conditions — Asthma | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Subjects took rosiglitazone 2 mg for 4 weeks, then 4mg for 4 weeks, then 8 mg for 4 weeks
  Interventions: Drug: rosiglitazone

INTERVENTIONS:
Drug: rosiglitazone — 2mg, 4mg, 8mg

SUMMARY:
Asthma is a common chronic disease characterized by airway inflammation and bronchoconstriction. This study utilizes the drug rosiglitazone (Avandia)to treat the effects of airway inflammation in patients with asthma.

The study will be conducted on 14 adult steroid naive patients with asthma. Patients with qualifying pulmonary function testing values will be eligible for enrollment. Enrolled subjects will be treated with rosiglitazone orally at 2mg dose for 4 weeks. Patients will be reassessed and dosing will increase in 4 week increments up to 8mg.

DETAILED DESCRIPTION:
The current standard-of-care utilizes corticosteroids to down-regulate the inflammatory state in patients with asthma. However, corticosteroids have many side effects and are not universally effective. New safe anti-inflammatory agents are needed to help modulate the disease. Peroxisome proliferator-activated receptor agonists are widely used to manage diabetes mellitus, another common chronic disease. These agents have been study models and have been shown to have anti-inflammatory effects in lung tissue. Case reports have noted improvement in asthma symptoms in patients being treated with these agents. These agents are ideally placed for human research given their long record of safe use in the treatment of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and grant a witnessed, written informed consent
* Must be greater than 19 years old
* Must be able to swallow a tablet
* Female participants must have a negative urine pregnancy test at visit 1 and throughout duration of the study
* Must have a history of physician diagnosed asthma
* Must have a baseline FEV1 >60% predicted
* Must be able to perform pulmonary function testing
* Must have methacholine-induced decrease in FEV1 of 20%
* Must be capable of withholding medications that may affect the methacholine challenge test
* Must be able to withstand a 30 day washout period for all inhaled corticosteroids
* Must be able to attend all office visits, 4 weeks apart for 12 weeks. Each visit will last approximately 2-3 hours

Exclusion Criteria:

* Age 18 or younger
* FEV1 <60% predicted value
* History or presence of significant renal, hepatic,neurologic, cardiovascular, hematologic, cerebrovascular, respiratory, endocrine, gastrointestinal, or collagen vascular disorder that in the Investigator's opinion could interfere with the study or require medical attention that would interfere with the study.
* History of cancer other than basal cell skin cancer
* History of hypoglycemia
* Current smokers, greater than 10 pack year history, or patients quitting less than 1 year prior to screening
* History within the past year of excessive alcohol intake or drug addiction
* History of respiratory infection requiring treatment with an antibiotic within 2 week prior to visit 1
* Chronic intermittent use of inhaled, oral, intra-muscular, topical or intravenous corticosteroids within 4 weeks of visit 1
* Inability to perform consistent spirometry or nitric oxide exhalation
* Treatment with an experimental, non-approved drug, or investigational drug within the past 30 days
* Known hypersensitivity to rosiglitazone
* History of noncompliance to medical regimens and participants who are considered to be potentially unreliable

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Wichman, MD, Principal Investigator — Creighton University Medical Center
Locations (1):
- Creighton University Medical Center, Department of Pulmonology and Critical Care, Omaha, Nebraska, United States

REFERENCES:
- [Background] Matsuura H, Adachi H, Smart RC, Xu X, Arata J, Jetten AM. Correlation between expression of peroxisome proliferator-activated receptor beta and squamous differentiation in epidermal and tracheobronchial epithelial cells. Mol Cell Endocrinol. 1999 Jan 25;147(1-2):85-92. doi: 10.1016/s0303-7207(98)00214-7. PMID 10195695
- [Background] Benayoun L, Letuve S, Druilhe A, Boczkowski J, Dombret MC, Mechighel P, Megret J, Leseche G, Aubier M, Pretolani M. Regulation of peroxisome proliferator-activated receptor gamma expression in human asthmatic airways: relationship with proliferation, apoptosis, and airway remodeling. Am J Respir Crit Care Med. 2001 Oct 15;164(8 Pt 1):1487-94. doi: 10.1164/ajrccm.164.8.2101070. PMID 11704601
- [Background] Woerly G, Honda K, Loyens M, Papin JP, Auwerx J, Staels B, Capron M, Dombrowicz D. Peroxisome proliferator-activated receptors alpha and gamma down-regulate allergic inflammation and eosinophil activation. J Exp Med. 2003 Aug 4;198(3):411-21. doi: 10.1084/jem.20021384. PMID 12900517
- [Background] Lee KS, Kim SR, Park SJ, Park HS, Min KH, Jin SM, Lee MK, Kim UH, Lee YC. Peroxisome proliferator activated receptor-gamma modulates reactive oxygen species generation and activation of nuclear factor-kappaB and hypoxia-inducible factor 1alpha in allergic airway disease of mice. J Allergy Clin Immunol. 2006 Jul;118(1):120-7. doi: 10.1016/j.jaci.2006.03.021. Epub 2006 May 19. PMID 16815147
- [Background] Hammad H, de Heer HJ, Soullie T, Angeli V, Trottein F, Hoogsteden HC, Lambrecht BN. Activation of peroxisome proliferator-activated receptor-gamma in dendritic cells inhibits the development of eosinophilic airway inflammation in a mouse model of asthma. Am J Pathol. 2004 Jan;164(1):263-71. doi: 10.1016/s0002-9440(10)63116-1. PMID 14695339
- [Background] Kim SR, Lee KS, Park HS, Park SJ, Min KH, Jin SM, Lee YC. Involvement of IL-10 in peroxisome proliferator-activated receptor gamma-mediated anti-inflammatory response in asthma. Mol Pharmacol. 2005 Dec;68(6):1568-75. doi: 10.1124/mol.105.017160. Epub 2005 Sep 8. PMID 16150927
- [Background] Honda K, Marquillies P, Capron M, Dombrowicz D. Peroxisome proliferator-activated receptor gamma is expressed in airways and inhibits features of airway remodeling in a mouse asthma model. J Allergy Clin Immunol. 2004 May;113(5):882-8. doi: 10.1016/j.jaci.2004.02.036. PMID 15131570
- [Background] Ward JE, Gould H, Harris T, Bonacci JV, Stewart AG. PPAR gamma ligands, 15-deoxy-delta12,14-prostaglandin J2 and rosiglitazone regulate human cultured airway smooth muscle proliferation through different mechanisms. Br J Pharmacol. 2004 Feb;141(3):517-25. doi: 10.1038/sj.bjp.0705630. Epub 2004 Jan 12. PMID 14718259
- [Background] Wang AC, Dai X, Luu B, Conrad DJ. Peroxisome proliferator-activated receptor-gamma regulates airway epithelial cell activation. Am J Respir Cell Mol Biol. 2001 Jun;24(6):688-93. doi: 10.1165/ajrcmb.24.6.4376. PMID 11415933
- [Background] Hashimoto Y, Nakahara K. Improvement of asthma after administration of pioglitazone. Diabetes Care. 2002 Feb;25(2):401. doi: 10.2337/diacare.25.2.401. No abstract available. PMID 11815521
- [Background] Kharitonov SA, Gonio F, Kelly C, Meah S, Barnes PJ. Reproducibility of exhaled nitric oxide measurements in healthy and asthmatic adults and children. Eur Respir J. 2003 Mar;21(3):433-8. doi: 10.1183/09031936.03.00066903a. PMID 12661997
- [Background] Eder W, Ege MJ, von Mutius E. The asthma epidemic. N Engl J Med. 2006 Nov 23;355(21):2226-35. doi: 10.1056/NEJMra054308. No abstract available. PMID 17124020

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was through pulmonary and allergy/immunology clinics from September 2008 to November 2009.
Pre-assignment Details: 32 patients assessed for eligibility. 16 did not meet inclusion criteria. None of the 16 participants allocated to treatment were excluded before the study began.
Groups:
- Rosiglitazone: Subjects will take rosiglitazone 2 mg for 4 weeks, then 4mg for 4 weeks, then 8 mg for 4 weeks
Period: Overall Study
Arm/Group | Rosiglitazone
Started | 16
Completed | 14
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rosiglitazone
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34 (24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Methacholine Responsiveness as Assessed by PC20,
Description: PC20 is the concentration of methacholine at which patients had a decrease in Forced Expiratory Volume in one second (FEV1) of 20%
Time Frame: patients were assessed at baseline and at 12 weeks
Population: 3 subjects were not included in the final analysis due to missing data. Two subjects withdrew by visit 3. 1 had missing data at visit 2 due to equipment failure.
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Rosiglitazone
Number analyzed (Participants) | 13
mg/mL
  Baseline | 3.27 (2.34)
  Week 12 | 8.71 (7.77)
Statistical Analysis 1: Comparison: Rosiglitazone; Test type: Superiority or Other; p = 0.048, ANOVA — Comparison is between baseline and week 12

2. Secondary Outcome: Exhaled Nitric Oxide in Parts Per Billion (Ppb), Parts Per Billion
Description: Fraction Exhaled Nitric oxide was measured on each visit prior to bronchoprovocation by chemiluminescence using an analyzer.
Time Frame: patients were assessed at baseline and 12 weeks
Population: 2 patients withdrew from the study in visit 3
Measure: Mean (Standard Deviation); unit: parts per billion
Arm/Group | Rosiglitazone
Number analyzed (Participants) | 14
parts per billion
  Baseline | 48 (32)
  12 weeks | 41 (35)
Statistical Analysis 1: Comparison: Rosiglitazone; Test type: Superiority or Other; p = 0.183, Friedman — comparison was at baseline and week 12; Mean Difference (Final Values) = 7, Standard Deviation 35

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 in liters
Time Frame: patients were assessed at baseline and 12 weeks
Population: Two subjects withdrew from the study in visit 3
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Rosiglitazone
Number analyzed (Participants) | 14
Liters
  Baseline | 2.95 (0.89)
  Week 12 | 3.04 (0.95)
Statistical Analysis 1: Comparison: Rosiglitazone; Test type: Superiority or Other; p = 0.398, Friedman — Comparison was at baseline and week 12; Mean Difference (Final Values) = 0.09, Standard Deviation 0.95

4. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Percent Predicted
Description: Spirometry was performed on each visit according to American Thoracic Society guidelines. FEV1 percent predicted was measured.
Time Frame: patients were assessed at baseline and 12 weeks
Population: Two subjects withdrew from the study in visit 3
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Rosiglitazone
Number analyzed (Participants) | 14
percent predicted
  Baseline | 82 (12)
  Week 12 | 85 (15)

ADVERSE EVENTS:
Arm/Group | Rosiglitazone
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
Small sample size. Lack of placebo control arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No